CLINICAL TRIAL: NCT03484988
Title: The Effect of n-3 PUFA Plant Oil Intake on Human Metabolism:A Randomized Double-Blind Trial
Brief Title: The Effect of n-3 PUFA Plant Oil Intake on Human Metabolism
Acronym: PUFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPG2017102074
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hyperlipidemias
Keywords: Polyunsaturated fatty acids; Echium oil; Hyperlipidemias; Metabolites; Gut Microbiota
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The all details of groups assignment are arranged and controlled by the research designers. The color, shape, and external packaging of the n-3 polyunsaturated fatty acid and placebo are consistent (faint yellow to yellow oil in transparent soft capsules). Each bottle of capsules will be marked with the name (or identify number) of the participants by research designers. Thus, the grouping of participants is blind to the rest of the researchers (like outcomes assessors).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo oil (Placebo Comparator): Ingredients: Corn oil, 500mg per capsule
  Interventions: Dietary Supplement: Placebo oil
- Echium oil (Experimental): Ingredients: Echium oil,500mg per capsule
  Interventions: Dietary Supplement: Echium oil
- Mixed oil (Experimental): Ingredients:Mixed oil(Echium oil,camelina oil,safflower oil) 500mg per capsule
  Interventions: Dietary Supplement: Mixed oil

INTERVENTIONS:
Dietary Supplement: Placebo oil — The participants were asked to take corn oil capsule twice a day, 4 capsules (500mg/capsules) each time. The intervention period is about 3 months. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Placebo oil
Dietary Supplement: Echium oil — The participants were asked to take echium oil capsule twice a day, 4 capsules (500mg/capsules) each time. The intervention period is about 3 months. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Echium oil
Dietary Supplement: Mixed oil — The participants were asked to take mixed oil(echium oil,camelina oil,safflower oil) twice a day, 4 capsules (500mg/capsules) each time. The intervention period is about 3 months. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Mixed oil

SUMMARY:
The findings of previous experiments suggested that polyunsaturated fatty acids(PUFAs) has been linked to anti-hyperlipidemia, and reducing the risk of cardiovascular disease.This is a randomized double-blind trial, aims to study the effect of PUFAs on blood lipids and human metabolism. Firstly, the investigators will investigate the efficacy of mixed plant oil(echium oil, camelina oil, safflower oil) and pure echium oil on improving the levels of blood lipids. Secondly, next generation sequencing (NGS), ultra-high performance liquid chromatography-tandem mass spectrometric (UPLC-MS/MS) and gas chromatography-mass spectrometry detection will be conducted to explore the role of PUFAs on gut microbiota as well as metabolites. Thirdly, single nucleotide polymorphism will be genotyped by Time-of-flight mass spectrometry to find the gene-environment interaction effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30-60 years of age
* Marginal elevated blood lipids or hyperlipidemia[Total cholesterol≥5.2 mmol/L(200 mg/dl) or triglyceride≥1.70 mmol/L(150mg/dl) or low density lipoprotein cholesterol≥3.4 mmol/L(130 mg/dl)]

Exclusion Criteria:

* Pregnancy；
* Known cardiovascular disease, diabetes, hypertension and any other chronic disease；
* Known gastrointestinal disease, such as Irritable Bowel Syndrome(IBS), functional bowel disease and so on；
* Acute or chronic inflammatory conditions;
* Liver or kidney dysfunction;
* An unwillingness to discontinue nutritional supplements；
* Use of lipid-lowering, antiinflammatory, antidepressant, or blood pressure medication;
* Evidence of drug or alcohol abuse；
* Take antibiotics or probiotics in the last three months.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes in blood lipids profile | At 0 week, 4th week, 12th week in intervention period
  Fasting serum total cholesterol, low density lipoprotein, high density lipoprotein and triglycerides
Changes in vascular inflammation markers | At 0 week, 4th week, 12th week in intervention period
  Fasting plasma C-reactive protein, soluble intercellular adhesion molecule-1, soluble vascular cell adhesion molecule-1, soluble E-selectin

SECONDARY OUTCOMES:
Changes in plasma metabolites | At 0 week, 4th week, 12th week in intervention period
  Plasma phospholipid fatty acid profile
Changes of microbiota metabolite in fecal | At 0 week, 4th week, 12th week in intervention period
  short chain fatty acids (SCFA)
Changes in gut microbiota | At 0 week, 4th week, 12th week in intervention period
  next generation sequencing
single nucleotide polymorphism genotype | At 0 week
  time of flight mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided